CLINICAL TRIAL: NCT03673696
Title: A Phase I, Single-center, Randomized，Double-blind, Placebo-controlled, Single & Multiple Ascending Dose Study to Assess the Tolerability and Pharmacokinetics of HEC74647PA Capsule in Healthy Adult Subjects
Brief Title: The Tolerability and Pharmacokinetics Study of HEC74647PA Capsule in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sunshine Lake Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HEC74647-P-01
Record Dates: First submitted 2018-09-10; First posted 2018-09-17 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2018-09

CONDITIONS: Chronic Hepatitis c
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- 50 mg single dose (Experimental): It includes two group, one group is pilot study, healthy subjects receive a single dose of 50 mg HEC74647PA capsule (N=2) . Another group is formal study, healthy subjects receive a single dose of 50 mg HEC74647PA capsule (N=8) or matching placebo (N=2).
  Interventions: Drug: HEC74647PA Capsule; Drug: placebo
- 100 mg single dose (Experimental): Healthy subjects, receiving a single dose of 100 mg HEC74647PA capsule (N=8) or matching placebo (N=2).
  Interventions: Drug: HEC74647PA Capsule; Drug: placebo
- 200 mg single dose (Experimental): Healthy subjects, receiving a single dose of 200 mg HEC74647PA capsule (N=16) or matching placebo (N=2) under fed or fasted conditions, this group is a two-sequence, two-period crossover study.
  Interventions: Drug: HEC74647PA Capsule; Drug: placebo
- 400 mg single dose (Experimental): Healthy subjects, receiving a single dose of 400 mg HEC74647PA capsule (N=8) or matching placebo (N=2).
  Interventions: Drug: HEC74647PA Capsule; Drug: placebo
- 600 mg single dose (Experimental): Healthy subjects, receiving a single dose of 600 mg HEC74647PA capsule (N=8) or matching placebo (N=2).
  Interventions: Drug: HEC74647PA Capsule; Drug: placebo
- 800 mg single dose (Experimental): Healthy subjects, receiving a single dose of 800 mg HEC74647PA capsule (N=8) or matching placebo (N=2).
  Interventions: Drug: HEC74647PA Capsule; Drug: placebo
- 100 mg multiple doses (Experimental): Healthy subjects, receiving 100 mg HEC74647PA capsule (N=10) or placebo(N=2) once daily (q.d.) for 7 days.
  Interventions: Drug: HEC74647PA Capsule; Drug: placebo
- 200 mg multiple doses (Experimental): Healthy subjects, receiving 200 mg HEC74647PA capsule (N=10) or placebo(N=2) once daily (q.d.) for 7 days.
  Interventions: Drug: HEC74647PA Capsule; Drug: placebo
- 400 mg multiple doses (Experimental): Healthy subjects, receiving 400 mg HEC74647PA capsule (N=10) or placebo(N=2) once daily (q.d.) for 7 days.
  Interventions: Drug: HEC74647PA Capsule; Drug: placebo

INTERVENTIONS:
Drug: HEC74647PA Capsule — Capsule administered orally once daily
Drug: placebo — Matching Placebo Capsule

SUMMARY:
The Tolerability and Pharmacokinetics Study of HEC74647PA Capsule in Healthy Adult Subjects

DETAILED DESCRIPTION:
A Phase I, Single Center, Randomized, Double-blind, Placebo-controlled, Single & Multiple Ascending Dose Study to Access the Tolerability and Pharmacokinetics of HEC74647PA Capsule in Healthy Adult Subjects.

ELIGIBILITY:
Inclusion Criteria:

* Able to comprehend and sign the ICF voluntarily prior to initiate the study;
* Able to complete the study according to the protocol;
* Between 18 and 45 years of age, inclusive, male subject should be no fertility needs;
* Body weight of male and female subject should be ≥50 kg and ≥45 kg respectively; Body Mass Index (BMI) is between 18 and 28 kg/m2, inclusive;
* Physical examination and vital signs without clinically significant abnormalities.

Exclusion Criteria:

* Smokers, who smoke more than 5 cigarettes/day within 3 months before the study;
* Drink frequently, namely alcohol consumption are 14 units per week (1 unit = 285 mL of beer, or 25 mL of strong wine, or 100 mL of grape wine);
* Donated blood or massive blood loss within 3 months before screening (>450 mL）;
* Have any disease that increases the risk of bleeding, such as acne, acute gastritis or stomach and duodenal ulcers;
* Have taken any prescription drug, over-the-counter drug, vitamin product or herbal medicine within 1 month prior to screening;
* Have participated in any clinical trial or taken any study drug within 3 months before dosing;
* Viral hepatitis（including CHB and CHC）and positive test result of anti-HIV Ab or syphilis.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 2018-09-04 (Actual); Primary Completion 2019-07-02 (Actual); Study Completion 2019-07-05 (Actual)

PRIMARY OUTCOMES:
Adverse events of the single ascending-dose | Baseline to day 6~13
  To assess the tolerability after a single dose of HEC74647PA capsule
Adverse events of the multiple ascending-dose | Baseline to day 12
  To assess the tolerability after multiple doses of HEC74647PA capsule
Tmax | Prior to dosing (0 h) and 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 36, 48, 72, 96 and 120 h after dosing
  Time of the maximum observed plasma concentration
AUC | Prior to dosing (0 h) and 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 36, 48, 72, 96 and 120 h after dosing
  Area under the plasma concentration-time curve (AUC)
Cmax | Prior to dosing (0 h) and 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 36, 48, 72, 96 and 120 h after dosing
  Maximum observed plasma concentration of HEC74647
T1/2 | Prior to dosing (0 h) and 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 36, 48, 72, 96 and 120 h after dosing
  Terminal elimination half-life
Vz/F | Prior to dosing (0 h) and 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 36, 48, 72, 96 and 120 h after dosing
  Apparent volume of distribution
CL/F | Prior to dosing (0 h) and 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 36, 48, 72, 96 and 120 h after dosing
  Oral clearance
MRT | Prior to dosing (0 h) and 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 36, 48, 72, 96 and 120 h after dosing
  Mean Residence Time

CONTACTS AND LOCATIONS:
Overall Officials: Yanhua Ding, Doctor, Principal Investigator — The First Hospital of Jilin University
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No